CLINICAL TRIAL: NCT03151369
Title: The Relationship Between Visual Pain Score and Perfusion Index in Postoperative Patients
Brief Title: Visual Pain Score and Perfusion Index in Postoperative Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assistant professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 17-KAEK-007
Record Dates: First submitted 2017-04-18; First posted 2017-05-12 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Perfusion
MeSH Terms: interventions — Morphine; Analgesics, Opioid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morphine (Other): patients with the visual analog scale over 3 will receive morphine
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — patients with the visual analog scale over 3 will receive morphine
  Other Names: opioid analgesic

SUMMARY:
The relationship between visual pain score and perfusion index in postoperative patients.

DETAILED DESCRIPTION:
The patients' operated with general anesthesia and who had visual pain score(VAS) above 3 will be measured postoperatively perfusion index. .If the VAS score is above 3, 2 mg of morphine will be made. When the VAS score is below 3, the perfusion index will be measured again.Thus, the changes between vas and perfusion index will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery with general anesthesia

Exclusion Criteria:

* Patients with caesarean section, pregnancy story and chronic pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Perfusion index Perfusion index | two times in one day
  Measurement of perfusion on the right ring finger

SECONDARY OUTCOMES:
visual analog scale | two times in one day
  measurement of pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Principal Investigator — Assistant professor
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided